CLINICAL TRIAL: NCT06512519
Title: A Multicenter Prospective Study of Second Haploidentical Transplantation for Graft Failure After the First Haploidentical Transplantation
Brief Title: Second Haplo-transplantation for Graft Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Ruijin Hospital (Other); Zhejiang University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Shandong Provincial Hospital (Other Government); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Fujian Medical University (Other); Hebei Yanda Ludaopei Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking University First Hospital (Other); Jiangsu Provincial People's Hospital (Other); Shengjing Hospital (Other); Xinqiao Hospital of Chongqing (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB181-001M
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Graft Failure; Stem Cell Transplant Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): second haploidentical stem cell transplantation
  Interventions: Other: second allogeneic stem cell transplantation

INTERVENTIONS:
Other: second allogeneic stem cell transplantation — 1. Change another donor if possible
  2. Conditioning regimen: fludarabine (30mg/m2/day, days -6 to -2 ), cyclophosphamide (1g/m2/day, days -5 to -4)
  3. GVHD prophylaxis: cyclosporine A (concentration 150-250ng/ml), mycophenolate mofetil (0.5g bid -3d to neutrophil engraftment)+anti CD25 monoAb (20mg -1d, +4d, +15d)

SUMMARY:
Graft failure is a fatal complication following allogeneic stem cell transplantation where a second transplantation is usually required for salvage. There are no recommended regimens for second transplantations for graft failure, especially in the haploidentical transplant setting. We recently reported encouraging outcomes using a novel method (haploidentical transplantation from a different donor after conditioning with fludarabine and cyclophosphamide). However, the study was performed in single-center and with very small sample size. Therefore, it should be further validated via multicenter study. In this multi-center study, we aim to further evaluate the safety and efficacy of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary disease: hematological malignancies (AML, CML, MDS, lymphoma, etc.); 2. Graft failure after the first haploidentical stem cell transplantation; 3. Time from the first transplantation to the second transplantation is less than 180 days; 4. Age≥14 years.

Exclusion Criteria:

* 1. Active infections; 2. Active GVHD; 3. Organ dysfunction: hepatic injury (Tbil≥2ULN), renal injury (Cr≥1.5ULN), heart injury (EF%<50% or symptomatic heart failure); 4. Eastern Cooperative Oncology Group (ECOG) score>2; 5. Expected life time<30 days; 5. Patients could not cooperate; 6. Other situations that are considered inappropriate for enrollment by the investigators,

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Engraftment of neutrophils | 28 days after second transplantation
  Engraftment of neutrophils was defined as the first of 3 consecutive days when the absolute neutrophil count achieved 500/uL.

SECONDARY OUTCOMES:
Engraftment of Platelet | 100 days after second transplantation
  Platelet engraftment was defined as the first of 7 consecutive days that platelet counts ≥20 × 10^9/L in the absence of platelet transfusion
TRM at 28 day | 28 days after second transplantation
  treatment-related mortality (TRM) was defined as death from any cause other than relapse
TRM at 100 day | 100 days after second transplantation
  treatment-related mortality (TRM) was defined as death from any cause other than relapse
GVHD | Participants will be followed for an expected average of 1 year
  Both acute and chronic GVHD was diagnosed and graded according to international criteria.
OS | Participants will be followed for an expected average of 1 year
  Overall survival (OS)
LFS | Participants will be followed for an expected average of 1 year
  Leukemia-free survival (LFS) was defined as the survival period with continuous CR.
CIR | Participants will be followed for an expected average of 1 year
  The cumulative incidence of relapse (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, M.D., Principal Investigator — Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No